CLINICAL TRIAL: NCT02366377
Title: An Efficacy, Safety, and Tolerability Study of SHR3824 in the Treatment of Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: The PK/PD, Efficacy, Safety and Tolerability Study of SHR3824 in Combination With Metformin in Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR3824-108
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — henagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- SHR3824 Placebo (Experimental): SHR3824 Placebo , once daily, 12 weeks, Metformin, Three times daily, 500mg, background drug.
  Interventions: Drug: Placebo; Drug: Metformin
- SHR3824 5 mg (Experimental): SHR3824 5 mg , once daily, 12 weeks, Metformin, Three times daily, 500mg, background drug.
  Interventions: Drug: SHR3824; Drug: Metformin
- SHR3824 10 mg (Experimental): SHR3824 10 mg , once daily, 12 weeks, Metformin, Three times daily, 500mg, background drug.
  Interventions: Drug: SHR3824; Drug: Metformin
- SHR3824 20 mg (Experimental): SHR3824 20mg , once daily, 12 weeks, Metformin, Three times daily, 500mg, background drug.
  Interventions: Drug: SHR3824; Drug: Metformin

INTERVENTIONS:
Drug: SHR3824
  Arms: SHR3824 10 mg; SHR3824 20 mg; SHR3824 5 mg
Drug: Placebo
  Arms: SHR3824 Placebo
Drug: Metformin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 3 different doses of SHR3824 compared with placebo in patients with type 2 diabetes mellitus who are receiving treatment with metformin monotherapy (ie, treatment with a single drug) and have inadequate glycemic (blood sugar) control.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of type 2 diabetes mellitus;
* Hemoglobin A1c levels >=7.5% and <=10.5%;
* Body mass index (BMI) 25 to 45 kg/m2;
* Patient either has been treated with metformin for more than 8 weeks with dose more than 1500mg/day.

Exclusion Criteria:

* Type I diabetes mellitus, diabetes mellitus resulting from pancreatic disorder, or secondary diabetes mellitus (acromegaly, Cushing's syndrome, etc.);
* Past or current history of severe diabetic complications (proliferative diabetic retinopathy, stage III or later stage overt nephropathy, diabetic ketoacidosis, or serious diabetic neuropathy);
* Systolic blood pressure of ≥160 mmHg or diastolic blood pressure of ≥100 mmHg on the start or end day of the run-in period;
* History of myocardial infarction, unstable angina, or cerebrovascular disorder within 6 months before the start of the run-in period;
* Past or current history of malignant tumor;
* Past or current history of drug hypersensitivity such as shock and anaphylactoid symptoms;
* Pregnant women, lactating mothers, or women of childbearing potential;
* Any condition that subjects are assessed to be ineligible by the investigator (sub investigator).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Adjusted Mean Change in HbA1c Levels | Baseline to Week 12
The number of volunteers with adverse events as a measure of safety and tolerability | Baseline to Week 12

SECONDARY OUTCOMES:
Adjusted Mean Change in Fasting Plasma Glucose | Baseline to Week 12
Proportion of Participants Achieving Glycemic Response Defined as HbA1c <7% | Baseline to Week 12